CLINICAL TRIAL: NCT02770547
Title: Leg Thermotherapy for Intermittent Claudication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601589496
Record Dates: First submitted 2016-05-05; First posted 2016-05-12 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Heat Thermotherapy (Active Comparator): Low heat thermotherapy will be applied to subject's leg. Subject will wear a garment through which heated water is circulated which in turn supplies low heat to the subject's leg.
  Interventions: Device: Low Heat Thermotherapy
- High Heat Thermotherapy (Experimental): High heat thermotherapy will be applied to subject's leg. Subject will wear a garment through which heated water is circulated which in turn supplies high heat to the subject's leg.
  Interventions: Device: High Heat Thermotherapy

INTERVENTIONS:
Device: Low Heat Thermotherapy — Subject will wear a High Density LCG (Liquid Circulating Garment). Water will be heated and circulated through the garment, which in turn supplies low heat to the subject's leg.
  Arms: Low Heat Thermotherapy
Device: High Heat Thermotherapy — Subject will wear a High Density LCG (Liquid Circulating Garment). Water will be heated and circulated through the garment, which in turn supplies high heat to the subject's leg.
  Arms: High Heat Thermotherapy

SUMMARY:
This study proposes to evaluate the potential of leg thermotherapy as a non-pharmacological intervention that could improve the mobility and exercise tolerance of patients with intermittent claudication. Thermotherapy is a simple, easily applicable therapy that enhances exercise tolerance in patients with chronic heart failure by improving peripheral vascular endothelial function.

DETAILED DESCRIPTION:
Peripheral arterial disease is characterized by atherosclerotic obstruction of the arteries in the lower extremities and affects approximately 10% of individuals older than 65 years. The most common clinical presentation of peripheral arterial disease is intermittent claudication, defined as leg pain caused by insufficient blood flow during walking. Individuals with intermittent claudication have severe exercise intolerance and markedly reduced levels of daily ambulatory activity. It is estimated that up to 40 million people worldwide suffer from intermittent claudication. Despite the increasing prevalence of this condition, few medical therapies improve mobility and exercise tolerance in these patients. An urgent need remains for the development of novel, non-invasive strategies that are more widely accessible and eliminate the need for supervision and frequent traveling to a clinical facility. The study proposes to evaluate the potential of leg thermotherapy as a non-pharmacological intervention that could improve the mobility and exercise tolerance of patients with intermittent claudication.

Subjects will complete baseline assessments for eligibility and ability to do study, including medical history, quality of life assessment, ankle-brachial measurement, leg MRI, venous blood draw, assessment of vascular function, and 6-minute walk test. Treatment consists of 3 treatment sessions per week for six consecutive weeks. Subjects will be randomized to low-heat therapy or high-heat therapy. Subjects will wear water-circulating pants through which the heat therapy will be administered during the treatment sessions. Outcome measurements (same as baseline assessments) will be repeated after 9 treatment sessions and after 18 treatment sessions (at the end of the treatment period).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a stable symptomatic claudication for ≥6 months
* Ankle brachial index <0.9

Exclusion Criteria:

* Uncontrolled Diabetes (HbA1C > 8.5 measured within 3 months prior to date of consent)
* Heart Failure
* Chronic Obstructive Pulmonary Disease
* Critical limb ischemia (ischemic rest pain or ischemia-related non healing wounds or tissue loss
* Prior amputation
* Exercise-limiting comorbidity (i.e., angina, chronic lung disease, or arthritis)
* Recent (<3 months) infrainguinal revascularization (surgery or endovascular revascularization) or revascularization planned during study period.
* Plans to change medical therapy during the duration of the study
* Active cancer
* Chronic kidney disease (eGFR <30 by Modification of Diet in Renal Disease or Mayo or Cockcroft-Gault formula).
* HIV positive, active hepatitis B virus (HBV) or hepatitis C virus (HCV) disease.
* Presence of any clinical condition that in the opinion of the principal investigator makes the patient not suitable to participate in the trial.
* Peripheral neuropathy, numbness, or paresthesia in the legs.
* Morbid obesity BMI > 35.
* Open wounds or ulcers on the extremity.

MRI Exclusions:

* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm clips
* Carotid artery vascular clamp
* Neurostimulator
* Insulin or infusion pump
* Implanted drug infusion device
* Bone growth/fusion stimulator
* Cochlear, otologic, or ear implant
* History of claustrophobia or who are unable to lie flat or who do not fit inside the bore of the scanner

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Tesini Roseguini, PhD, Study Director — Purdue University
Locations (2):
- United States (2):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Patient non-compliant | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.00 (7.80) | 68.73 (8.99) | 68.87 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 12 | 14 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Height [Mean (Standard Deviation); unit: cm] | 173.45 (7.09) | 175.20 (6.71) | 174.30 (6.84)
Weight [Mean (Standard Deviation); unit: kg] | 81.38 (15.83) | 85.67 (15.77) | 83.45 (15.67)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.93 (4.21) | 27.81 (4.11) | 27.36 (4.11)
Ankle-Brachial Index [Mean (Standard Deviation); unit: Ratio] — The ankle-brachial index represents the highest systolic pressure taken from the brachial artery divided by the highest systolic pressure obtained from the dorsalis pedis and posterior tibial arteries. This represents a ratio of upper limb blood pressure to lower limb blood pressure and is a hallmark diagnostic measure for peripheral artery disease.
  Ratio | 0.64 (0.11) | 0.70 (0.11) | 0.67 (0.11)
Number of Participants with Lower Limb Stents [Count of Participants; unit: Participants] | 6 | 7 | 13
Number of Participants with Type II Diabetes Mellitus [Count of Participants; unit: Participants] | 3 | 8 | 11
Smoker [Count of Participants; unit: Participants] | 7 | 6 | 13
6 minute walk test distance [Mean (Standard Deviation); unit: meters] | 386.38 (85.08) | 414.12 (109.23) | 400.25 (97.23)
Maximum absolute peak blood flow [Mean (Standard Deviation); unit: ml/s] — Population: Some MRI outputs were affected by technological problems and the data was subsequently removed from the final dataset. Addtionally, patients who could not undergo MRI due to non-compatible stenting or claustrophobia were also removed.
  ml/s
    number analyzed (Participants) | 7 | 7 | 14
    (all) | 3.87 (1.89) | 5.73 (3.30) | 4.80 (2.78)
Serum Endothelin-1 [Mean (Standard Deviation); unit: pg/ml] — Population: 1 participant could not under go blood draws and 1 participant's samples were deemed an outlier and subsequently removed.
  pg/ml
    number analyzed (Participants) | 14 | 14 | 28
    (all) | 2.44 (0.51) | 2.30 (0.49) | 2.37 (0.50)
Serum Total Nitrate [Mean (Standard Deviation); unit: uM] — Population: 1 participant could not under go blood draws.
  uM
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 64.32 (66.33) | 42.19 (25.74) | 53.64 (51.32)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 149.13 (12.45) | 153.54 (12.22) | 151.34 (12.33)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.82 (10.37) | 82.24 (8.85) | 81.53 (9.50)
Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 103.59 (9.83) | 106.01 (8.82) | 104.80 (9.26)
Cutaneous Vascular Conductance [Mean (Standard Deviation); unit: Percentage of maximum conductance] — Laser-Doppler flowmetry of skin included placement of two heating probes on the anterior portion of the lower leg. The participant sat in a semi-recumbent position for 70 minutes while the temperature of the probe progressed from 33C to 39C at minute 10 and then to 43C at minute 50. Cutaneous vascular conductance was calculated at the average red blood cell flux during the final 2 minutes of the 39C heating portion divided by the mean arterial pressure taken at that time.
  Percentage of maximum conductance | 51.91 (4.23) | 56.33 (2.78) | 54.12 (2.52)
SF-36 [Mean (Standard Deviation); unit: units on a scale] — All scales are scored 1-100, with 1 being the poorest rating and 100 being the most optimal.
  units on a scale
    Phyiscal Functioning | 45.00 (26.02) | 42.14 (16.14) | 43.57 (21.29)
    Role Physical | 45.09 (30.54) | 41.96 (21.01) | 43.53 (25.77)
    Bodily Pain | 49.57 (29.87) | 44.93 (14.98) | 47.17 (23.07)
    General Health | 54.81 (20.78) | 58.93 (17.85) | 56.94 (19.08)
    Vitality | 45.54 (26.34) | 50.83 (19.75) | 48.28 (22.90)
    Social Functioning | 67.86 (26.73) | 65.00 (26.81) | 66.38 (26.33)
    Role Emotional | 70.24 (31.98) | 60.71 (33.40) | 65.48 (32.45)
    Mental Health | 77.86 (17.40) | 72.00 (19.16) | 74.83 (18.25)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance Assessed by Measuring Distance (m) Walked in 6-minutes
Description: 6-minutes walk test
Time Frame: Maximal walking distances on a 6mwt were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: Included all participants that completed the study.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 15 | 15
meters
  Week 3 | 388.75 (85.08) | 414.96 (109.23)
  Week 6 | 404.29 (83.05) | 419.73 (113.83)

2. Primary Outcome: Blood Pressure
Description: Participants have systolic, diastolic and mean blood pressure recording 14 times during baseline, week 3 and week 6 experimental sessions.
Time Frame: Average blood pressure taken every 5 minutes for 70 minutes was obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: Includes all participants that completed the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 15 | 15
mmHg
  Systolic BP Week 3 | 146.29 (17.08) | 148.97 (12.51)
  Systolic BP Week 6 | 149.84 (9.61) | 150.21 (15.38)
  Diastolic BP Week 3 | 79.38 (10.74) | 79.72 (9.42)
  Diastolic BP Week 6 | 80.31 (8.98) | 81.44 (8.64)
  Mean Arterial Pressure Week 3 | 101.69 (12.18) | 102.81 (9.33)
  Mean Arterial Pressure Week 6 | 103.48 (7.90) | 104.36 (9.39)

3. Primary Outcome: Circulating Levels of Endothelin-1 (pg/mL)
Description: Blood draw
Time Frame: Serum endothelin-1 levels were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: One participant was excluded as an outlier from the low heat group. One participant in the high heat group did not have blood draws
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 14 | 14
pg/mL
  Endothelin-1 Week 3 | 2.44 (0.66) | 2.11 (0.37)
  Endothelin-1 Week 6 | 2.60 (0.69) | 2.00 (0.35)

4. Primary Outcome: Circulating Total Nitrate Levels (mmol)
Description: Blood Draw
Time Frame: Serum total nitrate levels were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 14 | 14
mmol
  Total Nitrate Levels Week 3 | 63.62 (30.60) | 47.61 (21.31)
  Total Nitrate Levels Week 6 | 58.31 (29.30) | 42.95 (19.57)

5. Secondary Outcome: Vascular Function Assessed by Leg MRI to Measure Peak Blood Flow in Popliteal Artery (ml/s)
Description: Phase contrast magnetic resonance imaging was performed on the leg that the patient indicated to have the most severe claudication. An inflation cuff was placed around the thigh and inflated to 75 mmHg above resting brachial systolic pressure for 5 minutes. After 5 minutes of inflation, the cuff was release and an additional 10 minutes of imaging took place.
Time Frame: Peak flows after post-occlusive reactive hyperemia were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 7 | 5
ml/s
  Week 3 | 4.25 (2.54) | 4.85 (1.94)
  Week 6 | 4.49 (2.51) | 5.49 (2.43)

6. Secondary Outcome: Vascular Function Measured by Ankle-brachial Index - Calculated by Dividing Higher of Posterior Tibial or Dorsalis Pedis Blood Pressure (mmHg) by Higher of Right or Left Arm Systolic Blood Pressure (mmHg)
Description: Ankle-brachial Index
Time Frame: Ankle-brachial index measures were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: Includes all participants that completed the study.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 15 | 15
ratio
  Week 3 | 0.64 (0.14) | 0.71 (0.13)
  Week 6 | 0.64 (0.12) | 0.71 (0.11)

7. Secondary Outcome: Vascular Function Measuring Leg Cutaneous Vascular Conductance - Measured by Laser-doppler Flowmetry of the Skin
Description: Laser-Doppler flowmetry of skin included placement of two heating probes on the anterior portion of the lower leg. The participant sat in a semi-recumbent position for 70 minutes while the temperature of the probe progressed from 33C to 39C at minute 10 and then to 43C at minute 50. Cutaneous vascular conductance was calculated at the average red blood cell flux during the final 2 minutes of the 39C heating portion divided by the mean arterial pressure taken at that time.
Time Frame: Maximal cutaneous vascular conductance values after 40 minutes of localized heating were obtained at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: Includes all participants that completed the study.
Measure: Mean (Standard Deviation); unit: percentage of maximum conductance
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 15 | 15
percentage of maximum conductance
  Week 3 | 55.08 (3.691) | 56.09 (4.892)
  Week 6 | 54.29 (4.077) | 52.66 (3.806)

8. Secondary Outcome: Patient Reported Functional Health and Well-being Using 36-item Short Form Health Survey
Description: 36-item Short Form Health Survey. All scales are scored 1-100, with 1 being the poorest rating and 100 being the most optimal.
Time Frame: SF-36 questionnaires were administered at weeks 3/6 and 6/6 of the study and compared to baseline values.
Population: Includes all participants that completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
Number analyzed (Participants) | 15 | 15
units on a scale
  Physical Functioning Week 3 | 48.08 (27.27) | 45.05 (16.59)
  Physical Functioning Week 6 | 42.67 (29.43) | 49.26 (20.20)
  Role Physical Week 3 | 50.00 (33.46) | 50.00 (24.55)
  Role Physical Week 6 | 50.42 (31.65) | 56.25 (28.84)
  Bodily Pain Week 3 | 45.85 (21.25) | 49.29 (20.60)
  Bodily Pain Week 6 | 50.33 (22.40) | 51.87 (18.28)
  General Health Week 3 | 54.92 (13.82) | 61.47 (20.20)
  General Health Week 6 | 55.33 (18.48) | 59.40 (21.67)
  Vitality Week 3 | 50.00 (21.95) | 52.08 (20.41)
  Vitality Week 6 | 55.00 (21.80) | 55.00 (22.19)
  Social Functioning Week 3 | 79.81 (30.85) | 75.00 (24.02)
  Social Functioning Week 6 | 75.83 (27.33) | 72.50 (24.64)
  Role Emotinoal Week 3 | 80.77 (27.51) | 65.00 (30.57)
  Role Emotional Week 6 | 71.67 (29.18) | 64.44 (30.12)
  Mental Health Week 3 | 81.92 (16.90) | 72.33 (16.99)
  Mental Health Week 6 | 79.67 (14.33) | 71.33 (22.71)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant over the course of 6 weeks of treatment.
Arm/Group | Low Heat Thermotherapy | High Heat Thermotherapy
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Heat Thermotherapy (N=16) | High Heat Thermotherapy (N=16)
Surface level burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Some PC-MRI data was unreliable or lost due to errors in the scanning HR monitor. Erroneous data sets were removed, which reduced the power for PC-MRI flow-related variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02770547/SAP_000.pdf
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT02770547/Prot_001.pdf